CLINICAL TRIAL: NCT03238833
Title: Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital
Brief Title: Poor Ovarian Responders Undergoing IVF Using Luteal Ovarian Stimulation Versus Follicular Ovarian Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS15-CT11-12
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Fertilization in Vitro
Keywords: In vitro fertilization; Poor ovarian responder; Luteal ovarian stimulation; Antagonist protocol; Cumulus cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- luteal ovarian stimulation (Experimental): The controlled ovarian stimulation in in vitro fertilization cycle was started since luteal phase.
  Interventions: Other: luteal ovarian stimulation
- follicular ovarian stimulation (Active Comparator): The controlled ovarian stimulation in in vitro fertilization cycle was started since early follicular phase phase.
  Interventions: Other: follicular ovarian stimulation

INTERVENTIONS:
Other: luteal ovarian stimulation — In the in vitro fertilization cycle, controlled ovarian stimulation was started since the luteal phase.
  Arms: luteal ovarian stimulation
Other: follicular ovarian stimulation — In the in vitro fertilization cycle, controlled ovarian stimulation was started since the follicular phase.
  Arms: follicular ovarian stimulation

SUMMARY:
The investigators attempted to compare the clinical outcomes and cumulus genes expression in poor ovarian responders undergoing luteal ovarian stimulation or follicular ovarian stimulation in in vitro fertilization cycles.

DETAILED DESCRIPTION:
Multiple follicular wave theory proposed by Baerwald et al. implied that follicle recruitment may occur in the luteal phase of menstrual cycle. Therefore, luteal phase ovarian stimulation (LPOS) was considered as a potential feasible stimulation method during in vitro fertilization (IVF) cycle. In the beginning, in order to avoid delaying cancer treatment, LPOS was applied for fertility preservation of cancer patients, showing no difference in numbers of oocyte retrieved, mature oocytes and fertilization rate between luteal or follicular phase stimulation. In the recent, LPOS was used for infertility women, suggesting that LPOS owned quite good IVF outcomes. In previous studies, premature luteinizing hormone (LH) surge, a major reason worsening ovarian quality in poor ovarian responders (PORs), was seldom found in LPOS. High progesterone in luteal phase may aid in suppressing premature LH surge. An updated research claimed that numbers of oocyte retrieved, mature oocytes and fertilized oocytes in LPOS significantly increased when compared to follicular ovarian stimulation. Therefore, the investigators presumed that LPOS was a more effective method than follicular stimulation in PORs.

ELIGIBILITY:
Inclusion Criteria:

* Poor ovarian responders (PORs) met the Bologna criteria, having at least two of the three following features:

  1. advanced maternal age (≥ 40 years) or any other risk factor for POR,
  2. a previous POR (≤ 3 oocytes with a conventional stimulation protocol), and
  3. an abnormal ovarian reserve test. An abnormal ovarian reserve test was defined as antral follicle count (AFC) < 5 or anti-Müllerian hormone (AMH) < 1 ng/mL in this study.

Moreover, two episodes of a previous POR after maximal stimulation alone would be sufficient to define a patient as a POR.

Exclusion Criteria:

* oophorectomy
* exposure to cytotoxic or pelvic irradiation for malignancy
* taking herbal drugs or other hormonal agents

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
oocytes and embryos | through study completion, an average of 1 year
  retrieved oocytes in number, matured oocytes in number, fertilized oocytes in number, day 3 embryos in number, top-quality day 3 embryos in number

SECONDARY OUTCOMES:
pregnancy rate | Pregnancy will be confirmed 4 weeks after embryo transfer.
  Clinical pregnancy rate
genes expression | through study completion, an average of 1 year
  cumulus cells genes expression

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, PhD, Study Director — Kaohsiung Veterans General Hospital.; Salvatore Giovanni Vitale, M.D., Principal Investigator — University of Messina
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Baerwald AR, Adams GP, Pierson RA. Ovarian antral folliculogenesis during the human menstrual cycle: a review. Hum Reprod Update. 2012 Jan-Feb;18(1):73-91. doi: 10.1093/humupd/dmr039. Epub 2011 Nov 8. PMID 22068695
- [Result] Bedoschi GM, de Albuquerque FO, Ferriani RA, Navarro PA. Ovarian stimulation during the luteal phase for fertility preservation of cancer patients: case reports and review of the literature. J Assist Reprod Genet. 2010 Aug;27(8):491-4. doi: 10.1007/s10815-010-9429-0. Epub 2010 May 9. PMID 20455017
- [Result] von Wolff M, Thaler CJ, Frambach T, Zeeb C, Lawrenz B, Popovici RM, Strowitzki T. Ovarian stimulation to cryopreserve fertilized oocytes in cancer patients can be started in the luteal phase. Fertil Steril. 2009 Oct;92(4):1360-1365. doi: 10.1016/j.fertnstert.2008.08.011. Epub 2008 Oct 18. PMID 18930226
- [Result] Maman E, Meirow D, Brengauz M, Raanani H, Dor J, Hourvitz A. Luteal phase oocyte retrieval and in vitro maturation is an optional procedure for urgent fertility preservation. Fertil Steril. 2011 Jan;95(1):64-7. doi: 10.1016/j.fertnstert.2010.06.064. Epub 2010 Aug 5. PMID 20688325
- [Result] Cakmak H, Rosen MP. Ovarian stimulation in cancer patients. Fertil Steril. 2013 May;99(6):1476-84. doi: 10.1016/j.fertnstert.2013.03.029. PMID 23635348
- [Result] Cakmak H, Katz A, Cedars MI, Rosen MP. Effective method for emergency fertility preservation: random-start controlled ovarian stimulation. Fertil Steril. 2013 Dec;100(6):1673-80. doi: 10.1016/j.fertnstert.2013.07.1992. Epub 2013 Aug 26. PMID 23987516
- [Result] Kuang Y, Hong Q, Chen Q, Lyu Q, Ai A, Fu Y, Shoham Z. Luteal-phase ovarian stimulation is feasible for producing competent oocytes in women undergoing in vitro fertilization/intracytoplasmic sperm injection treatment, with optimal pregnancy outcomes in frozen-thawed embryo transfer cycles. Fertil Steril. 2014 Jan;101(1):105-11. doi: 10.1016/j.fertnstert.2013.09.007. Epub 2013 Oct 23. PMID 24161646
- [Result] Martinez F, Clua E, Devesa M, Rodriguez I, Arroyo G, Gonzalez C, Sole M, Tur R, Coroleu B, Barri PN. Comparison of starting ovarian stimulation on day 2 versus day 15 of the menstrual cycle in the same oocyte donor and pregnancy rates among the corresponding recipients of vitrified oocytes. Fertil Steril. 2014 Nov;102(5):1307-11. doi: 10.1016/j.fertnstert.2014.07.741. Epub 2014 Aug 22. PMID 25154677
- [Result] Kuang Y, Chen Q, Hong Q, Lyu Q, Ai A, Fu Y, Shoham Z. Double stimulations during the follicular and luteal phases of poor responders in IVF/ICSI programmes (Shanghai protocol). Reprod Biomed Online. 2014 Dec;29(6):684-91. doi: 10.1016/j.rbmo.2014.08.009. Epub 2014 Sep 6. PMID 25444501
- [Result] Li Y, Yang W, Chen X, Li L, Zhang Q, Yang D. Comparison between follicular stimulation and luteal stimulation protocols with clomiphene and HMG in women with poor ovarian response. Gynecol Endocrinol. 2016;32(1):74-7. doi: 10.3109/09513590.2015.1081683. Epub 2015 Sep 15. PMID 26370530
- [Result] Wei LH, Ma WH, Tang N, Wei JH. Luteal-phase ovarian stimulation is a feasible method for poor ovarian responders undergoing in vitro fertilization/intracytoplasmic sperm injection-embryo transfer treatment compared to a GnRH antagonist protocol: A retrospective study. Taiwan J Obstet Gynecol. 2016 Feb;55(1):50-4. doi: 10.1016/j.tjog.2015.07.001. PMID 26927248
- [Derived] Chen YC, Li JY, Li CJ, Tsui KH, Wang PH, Wen ZH, Lin LT. Luteal Phase Ovarian Stimulation versus Follicular Phase Ovarian Stimulation results in different Human Cumulus cell genes expression: A pilot study. Int J Med Sci. 2021 Feb 4;18(7):1600-1608. doi: 10.7150/ijms.55955. eCollection 2021. PMID 33746576
- [Derived] Lin LT, Vitale SG, Chen SN, Wen ZH, Tsai HW, Chern CU, Tsui KH. Luteal Phase Ovarian Stimulation May Improve Oocyte Retrieval and Oocyte Quality in Poor Ovarian Responders Undergoing In Vitro Fertilization: Preliminary Results from a Single-Center Prospective Pilot Study. Adv Ther. 2018 Jun;35(6):847-856. doi: 10.1007/s12325-018-0713-1. Epub 2018 Jun 4. PMID 29869107